CLINICAL TRIAL: NCT05474157
Title: Sarcopenia and Related Factors in COVID-19 Following Intensive Care
Brief Title: Sarcopenia and Related Factors in Coronavirus Disease 2019 (COVID-19) Following Intensive Care
Status: Terminated | Type: Observational
Why Stopped: techincal reasons
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.221.IRB1.071
Record Dates: First submitted 2020-12-07; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2020-12

CONDITIONS: Sarcopenia; Covid19; Intensive Care Unit Acquired Weakness
Keywords: Sarcopenia; covid19; acute respiratory distress syndrome; intensive care unit
MeSH Terms: conditions — Sarcopenia; COVID-19; Respiratory Distress Syndrome | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 15 patients Patients followed in the Intensive Care Unit due to COVID-19 infection
  Interventions: Other: Standard care treatment for COVID-19 in Intensive Care Unit
- Control group: 15 patients Patients who admitted to the 'Physical Medicine and Rehabilitation' clinic for other reasons during the pandemic period

INTERVENTIONS:
Other: Standard care treatment for COVID-19 in Intensive Care Unit — Standard care for ARDS patients consisted of respiratory support, intravenous fluid therapy, medical treatment including anticoagulation and sedation, nutrition, change of position every 4 hours and if needed, hemodynamic support.
  Groups: Study group

SUMMARY:
The primary aim of this study is to evaluate the patients who had pneumonia or severe acute respiratory distress syndrome (ARDS) due to COVID-19 in terms of sarcopenia and related factors following Intensive Care Unit (ICU).

The patients who had COVID-19 infection in the ICU and the patients who admitted to the 'Physical Medicine and Rehabilitation' clinic for other reasons during the pandemic period will be compared in terms of sarcopenia.

DETAILED DESCRIPTION:
Patients with acute respiratory distress syndrome (ARDS) could develop muscle weakness associated with impairment of physical function defined as intensive care unit acquired weakness. Significant muscle loss occurs in the first week of the Intensive Care Unit (ICU) hospitalizations due to acute respiratory failure. Patients lose 18 percent of their body weight when discharged from the ICU. The presence of sepsis is known as the hypercatabolic process for the muscles. Hypophosphatemia and hypomagnesemia can cause respiratory muscle weakness. Fever and inflammation, use of muscle relaxant or sedatives may also cause muscle loss in intensive care during this period.

COVID-19 is an acute infection with a high risk of enormous cytokine storm exacerbating the clinical condition in acute respiratory distress syndrome and is thought to further increase the risk of muscle weakness.

The patients will be evaluated for hand grip strength, calf circumference measurement, 'Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls' (SARCF), SarQoL, timed up and go test, sit to stand test, and Short form-36.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ARDS or severe pneumonia due to COVID-19 hospitalized in intensive care unit
* > 18 years old
* Age and gender matched patients admitted to the 'Physical Medicine and Rehabilitation' clinic for control group

Exclusion Criteria:

* Other diseases that may cause sarcopenia (cancer, non-respiratory organ failure and heart, liver or kidney failure)
* Neurological diseases that may cause sarcopenia (stroke, spinal cord injury, muscle diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with ARDS or severe pneumonia due to COVID-19 hospitalized in intensive care unit, >18 years Study group: 15 Control group: 15
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 12 months
  Hand grip strength is an indicator of overall muscle strength that predicts mortality in older patients. Hand grip strength was measured using a handheld dynamometer according to the instructions of the American Society of Hand Therapists.Patients were seated placing their arms by their sides with the elbow flexed to 90°, the forearm mid-prone, and the wrist in neutral position. Patients were asked to grip the dynamometer with maximal effort using standard verbal encouragement. Three trials were performed in the dominant hand with a 30 sec rest between trials and the highest value was recorded in kg. The cut-off values of grip strength is 28.6 kg in men and 16.4 kg in women.

SECONDARY OUTCOMES:
Calf circumference measurement | 12 months
  Calf circumference which positively correlate with appendicular skeletal muscle mass could be used as a surrogate tool of muscle mass for sarcopenia. Adding calf circumference to SARC-F significantly improves the sensitivity and overall diagnostic accuracy of SARC-F in Chinese community dwelling older adults. Calf circumference of the patients was measured while patients in supine position, with left knee raised and calf at right angles to the thigh, using flexible plastic tape at the greatest circumference without compression of the subcutaneous tissue. The measurement were repeated 2 times and average value was recorded. According to 'European Working Group on Sarcopenia in Older People', calf circumference measure on the left leg for right-handed persons in a sitting position with the knee and ankle at a right angle and feet resting on the floor so we measured the left side for sarcopenia.
SARC-F (Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls) | 12 months
  To evaluate sarcopenia SARC-F was applied as a screening questionnaire. It is a self-filled survey questionnaire consisting of five items. The most commonly used criteria for sarcopenia in clinical practice are 'European Working Group on Sarcopenia in Older People' (EWGSOP). EWGSOP recommends using the SARC-F test for risk assessment in patients at risk of sarcopenia. Turkish validation study of the test has been done.
Sit to stand test | 12 months
  Sit to stand test was used to evaluate strength and endurance of lower limbs. Patients are asked to sit on a chair by crossing their hands over their chest. They are asked to sit five times consecutively as fast as possible. The test is started in the sitting position and the test is terminated at the last standing position and the time is recorded. The test is carried out 2 times and the best grade obtained is recorded
Timed up and go test | 12 months
  To assess physical function/performance, timed up and go test was performed. It is an objective, reliable and simple test to evaluate balance and functional movement. The patient is asked to get up from a chair, walk 3 m, turn around, walk back and sit on the chair again. The time is recorded in how many seconds the patient has finished the test. The test is started and ended when the patient sit on the chair with back supported. It predicts mortality
Sarcopenia Quality of Life (SarQoL ) | 12 months
  To evaluate the impact of sarcopenia on quality of life SarQoL was administered. This test identifies and predicts sarcopenia complications that can affect the patient's quality of life. It helps to evaluate the patient's perception of their health, physical, psychological and social aspects to healthcare professional. SarQoL has been found reliable for use in clinical care and research study
Short form - 36 | 12 months
  Short form - 36 measures health related quality of life. It is a self-reported survey that evaluates individual health status with eight parameters consisting of physical function, pain, role limitations attributed to physical problems, role limitations attributed to emotional problems, mental health, social functioning, energy/ vitality, general health perception. There is not a summary score, each section is scored between 0-100, 0 indicates the worst condition, 100 indicates the best.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data

REFERENCES:
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Result] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Result] Gerovasili V, Stefanidis K, Vitzilaios K, Karatzanos E, Politis P, Koroneos A, Chatzimichail A, Routsi C, Roussos C, Nanas S. Electrical muscle stimulation preserves the muscle mass of critically ill patients: a randomized study. Crit Care. 2009;13(5):R161. doi: 10.1186/cc8123. Epub 2009 Oct 8. PMID 19814793
- [Result] Rantanen T, Volpato S, Ferrucci L, Heikkinen E, Fried LP, Guralnik JM. Handgrip strength and cause-specific and total mortality in older disabled women: exploring the mechanism. J Am Geriatr Soc. 2003 May;51(5):636-41. doi: 10.1034/j.1600-0579.2003.00207.x. PMID 12752838
- [Result] Turan Z, Ozyemisci Taskiran O, Erden Z, Kokturk N, Kaymak Karatas G. Does hand grip strength decrease in chronic obstructive pulmonary disease exacerbation? A cross-sectional study. Turk J Med Sci. 2019 Jun 18;49(3):802-808. doi: 10.3906/sag-1811-22. PMID 31190519
- [Result] Yoo JI, Choi H, Ha YC. Mean Hand Grip Strength and Cut-off Value for Sarcopenia in Korean Adults Using KNHANES VI. J Korean Med Sci. 2017 May;32(5):868-872. doi: 10.3346/jkms.2017.32.5.868. PMID 28378563
- [Result] Kawakami R, Murakami H, Sanada K, Tanaka N, Sawada SS, Tabata I, Higuchi M, Miyachi M. Calf circumference as a surrogate marker of muscle mass for diagnosing sarcopenia in Japanese men and women. Geriatr Gerontol Int. 2015 Aug;15(8):969-76. doi: 10.1111/ggi.12377. Epub 2014 Sep 20. PMID 25243821
- [Result] Yang M, Hu X, Xie L, Zhang L, Zhou J, Lin J, Wang Y, Li Y, Han Z, Zhang D, Zuo Y, Li Y, Wu L. Screening Sarcopenia in Community-Dwelling Older Adults: SARC-F vs SARC-F Combined With Calf Circumference (SARC-CalF). J Am Med Dir Assoc. 2018 Mar;19(3):277.e1-277.e8. doi: 10.1016/j.jamda.2017.12.016. PMID 29477774
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Bahat G, Oren MM, Yilmaz O, Kilic C, Aydin K, Karan MA. Comparing SARC-F with SARC-CalF to Screen Sarcopenia in Community Living Older Adults. J Nutr Health Aging. 2018;22(9):1034-1038. doi: 10.1007/s12603-018-1072-y. PMID 30379299
- [Result] Beaudart C, McCloskey E, Bruyere O, Cesari M, Rolland Y, Rizzoli R, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Bautmans I, Bertiere MC, Brandi ML, Al-Daghri NM, Burlet N, Cavalier E, Cerreta F, Cherubini A, Fielding R, Gielen E, Landi F, Petermans J, Reginster JY, Visser M, Kanis J, Cooper C. Sarcopenia in daily practice: assessment and management. BMC Geriatr. 2016 Oct 5;16(1):170. doi: 10.1186/s12877-016-0349-4. PMID 27716195
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Dardenne N, Bruyere O. Validation of the SarQoL(R), a specific health-related quality of life questionnaire for Sarcopenia. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):238-244. doi: 10.1002/jcsm.12149. Epub 2016 Oct 22. PMID 27897430
- [Result] Dodoo-Schittko F, Brandstetter S, Blecha S, Thomann-Hackner K, Brandl M, Knuttel H, Bein T, Apfelbacher C. Determinants of Quality of Life and Return to Work Following Acute Respiratory Distress Syndrome. Dtsch Arztebl Int. 2017 Feb 17;114(7):103-109. doi: 10.3238/arztebl.2017.0103. PMID 28302253